CLINICAL TRIAL: NCT03951220
Title: The Development and Pilot Testing of a New Magnetic Resonance (MR) Imaging Protocol to Quantify Both Myeloma Disease Burden and Associated Bone Loss
Brief Title: The Development and Pilot Testing of a New MR Imaging Protocol to Quantify Myeloma Disease Burden and Bone Loss
Acronym: LOOMIS
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Karthik Ramasamy, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 12548
Record Dates: First submitted 2019-05-01; First posted 2019-05-15 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Myeloma; Monoclonal Gammopathy of Undetermined Significance (MGUS); Smouldering Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell; Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma | interventions — Absorptiometry, Photon; Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloods and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1- Myeloma: Participants will be recruited at the point of either diagnosis or relapse. Any standard investigations that the clinician deems necessary will be carried out. Following recruitment, participants will undergo the first study appointment, the experimental combined MR imaging protocol, the DXA imaging scan and the bone biomarker blood and urine tests.
  This will be repeated at 6 months.
  Interventions: Other: Diffusion Weighted Magnetic Resonance Imaging (DWMRI); Other: DXA scan; Other: Bloods and urine
- Group 2- MGUS: Participants will be recruited at the point of either diagnosis or relapse. Any standard investigations that the clinician deems necessary will be carried out. Following recruitment, participants will undergo the first study appointment, the experimental combined MR imaging protocol, the DXA imaging scan and the bone biomarker blood and urine tests.
  This will be repeated at 6 months.
  Interventions: Other: Diffusion Weighted Magnetic Resonance Imaging (DWMRI); Other: DXA scan; Other: Bloods and urine
- Group 3- Healthy Volunteers: Participants will have the experimental combined MR imaging.
  Interventions: Other: Diffusion Weighted Magnetic Resonance Imaging (DWMRI)

INTERVENTIONS:
Other: Diffusion Weighted Magnetic Resonance Imaging (DWMRI) — Using the expertise of the Oxford Centre For Clinical Magnetic Resonance Research (OCMR) for imaging protocol development, and the new Fine Structural Analysis (FSA, Osteotronix Ltd, formerly Acuitas Medical) bone density quantification MRI method (Rafferty et al 2016), we will test a single protocol which combines three emerging experimental imaging sequences into a simple, non-invasive whole body imaging protocol to quantify disease burden and bone disease. To our knowledge, this has never been done before; if shown to be feasible, such a method would have two important applications: to precisely guide commissioned therapies in the clinic, so improving patient management; and as an exciting, novel research tool for the longitudinal combined assessment of tumour burden and cancer-induced bone disease in response to therapy.
Other: DXA scan — Used to assess bone density
  Groups: Group 1- Myeloma; Group 2- MGUS
Other: Bloods and urine — Samples will be taken to assess bone biomarkers
  Groups: Group 1- Myeloma; Group 2- MGUS

SUMMARY:
In the proposed study, the investigators will aim to develop and pilot a Magnetic Resonance (MR) imaging protocol and assess its ability to achieve the following: quantification of tumour burden and bone loss, detecting longitudinal changes in tumour load with therapy and detecting longitudinal changes in microarchitecture with therapy. The investigators also aim to investigate whether bone loss is better, worse or the same with different imaging techniques. This will be investigated by correlating the DXA imaging data with Diffusion-Weighted Magnetic Resonance Imaging (DWMRI) to see if it is possible to achieve quantifiable data of bone density.

DETAILED DESCRIPTION:
In the proposed study, the investigators will aim to develop and pilot a Magnetic Resonance (MR) imaging protocol and assess its ability to achieve the following: quantification of tumour burden and bone loss, detecting longitudinal changes in tumour load with therapy and detecting longitudinal changes in microarchitecture with therapy. The investigators also aim to investigate whether bone loss is better, worse or the same with different imaging techniques. This will be investigated by correlating the DXA imaging data with Diffusion-Weighted Magnetic Resonance Imaging (DWMRI) to see if it is possible to achieve quantifiable data of bone density.

Using the expertise of the Oxford Centre For Clinical Magnetic Resonance Research (OCMR) for imaging protocol development, and the new Fine Structural Analysis (FSA, Osteotronix Ltd, formerly Acuitas Medical) bone density quantification MRI method (Rafferty et al 2016), the investigators will test a single protocol which combines three emerging experimental imaging sequences into a simple, non-invasive whole body imaging protocol to quantify disease burden and bone disease. This has never been done before; if shown to be feasible, such a method would have two important applications: to precisely guide commissioned therapies in the clinic, so improving patient management; and as an exciting, novel research tool for the longitudinal combined assessment of tumour burden and cancer-induced bone disease in response to therapy.

The investigators hypothesize that this imaging tool will be superior to the combined current standard-of-care investigations in the quantification of tumour burden and bone loss. There are currently no tools available for quantifying structural changes to bone and overall bone loss in myeloma.

ELIGIBILITY:
Inclusion Criteria (All Groups):

* Participant is able to and willing to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.

Inclusion Criteria (Groups 1 and 2):

* Newly diagnosed myeloma or newly relapsed myeloma eligible for next therapy.
* Smouldering myeloma or intermediate or high risk MGUS.
* Patients attending Oxford NHS Haematology-Oncology centre.
* Diagnoses of MGUS, Smouldering Myeloma and MM made in accordance with the clinical diagnostic criteria set forth by IMWG (International Myeloma Working Group).

Exclusion Criteria (All Groups):

* Those who are unable or unwilling to give informed consent.
* Women who may be pregnant, breast feeding or women of child-bearing potential who are unwilling or unable to take sufficient precautionary measures will be excluded due to DXA imaging.

Exclusion Criteria (Groups 1 and 2):

* Signs of Spinal Cord Compression.
* Patients with documented metastatic lesions from another type of malignancy.
* Known contraindication for a MRI scan, including unacceptable pain on lying flat for 1 hour.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in Groups 1 & 2 will be recruited via the Haematology Outpatients clinic in Churchill Hospital.
  Group 3 participants will be recruited from the community
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ramasamy, Principal Investigator — University of Oxford Hospitals NHS Foundation Trust
Locations (1):
- Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from Groups 1 and 2 were identified and approached by a healthcare professional in the oncology clinic at the Churchill Hospital, Oxford. Group 3 participants were typically partners of the participants from Groups 1 and 2 and were recruited at the same time.
Groups:
- Group 1- Myeloma: Group 1a: New Myeloma; Group 1b: Relapsed Myeloma Group;1c: Smouldering Myeloma
  Baseline AND Follow-Up Assessment:
  Novel MR Whole body DXA scan Blood and urine samples QOL & scan experience questionnaires
- Group 2- MGUS: Baseline AND Follow-Up Assessment:
  Novel MR Whole body DXA scan Blood and urine samples QOL & scan experience questionnaires
- Group 3- Healthy Volunteers: Baseline Assessment ONLY:
  * Novel MR
  * QOL & scan experience questionnaires
Period: Overall Study
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers
Started (Enrolment) | 41 | 14 | 12
Baseline Assessment (GROUP 1 & 2 ASSESSMENT * Experimental MR * Whole body DXA scan * Blood and urine samples * QOL & scan experience questionnaires GROUP 3 ASSESSMENT * Experimental MR * QOL & scan experience questionnaires) | 41 | 14 | 12
Follow-Up Assessment (GROUP 1 & 2 ASSESSMENT * Experimental MR * Whole body DXA scan * Blood and urine samples * QOL & scan experience questionnaires GROUP 3 ASSESSMENT • (No follow-up)) | 32 | 12 | 0 (Group 3 participants did not attend follow-up)
Completed | 32 | 12 | 12
Not Completed | 9 | 2 | 0
Not completed — Withdrawal by Subject | 9 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Total 67 participants: Group 1a (new myeloma = 14), Group 1b (relapsed myeloma = 12), Group 1c (smouldering myeloma = 15), Group 2 (MGUS = 14), Group 3 (healthy volunteer = 12)
Groups:
- Group 1- Myeloma: Group 1a: New Myeloma Group 1b: Relapsed Myeloma Group 1c: Smouldering Myeloma
  Baseline AND Follow-Up Assessment:
  * Novel MR
  * Whole body DXA scan
  * Blood and urine samples
  * QOL & scan experience questionnaires
- Group 2- MGUS: Baseline AND Follow-Up Assessment:
  * Novel MR
  * Whole body DXA scan
  * Blood and urine samples
  * QOL & scan experience questionnaires
- Total: Total of all reporting groups
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers | Total
Number analyzed (Participants) | 41 | 14 | 12 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 7 | 7 | 31
  >=65 years | 24 | 7 | 5 | 36
Age, Continuous [Median (Full Range); unit: years] | 67.7 [40.9 to 85.3] | 65.5 [54.3 to 82.3] | 60.5 [35.2 to 75.5] | 65.6 [35.2 to 85.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 5 | 23
  Male | 30 | 7 | 7 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 41 | 14 | 12 | 67

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome 1: Quantifying Tumour Burden [Correlations With Apparent Diffusion Coefficient (ADC) Measurements]
Description: Primary Objective 1: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone biomarkers can improve quantification of tumour burden in patients with new or relapsed myeloma at baseline assessment, compared to paraprotein levels alone.
  This particular section analysed the correlation between the Apparent Diffusion Coefficient (ADC) measurements (from the Diffusion Weighted Magnetic Resonance Imaging (DW-MRI) component of the sequences) of lytic bone lesions, with standard clinical correlates of tumour burden (serum paraprotein, and serum paraprotein-associated immunoglobulin level).
  The measurement of ADC from DW-MRI is further described by Messiou et. al. [1]
  [1] Messiou, Christina, et al. "Guidelines for acquisition, interpretation, and reporting of whole-body MRI in myeloma: myeloma response assessment and diagnosis system (MY-RADS)." Radiology 291.1 (2019): 5-13.
Time Frame: At baseline
Population: Subset of Group 1a and 1b, on active chemotherapy, with lytic bone lesions identified on baseline novel MR scan, amenable to ADC measurement, and a paired baseline serum paraprotein, or paraprotein-associated immunoglobulin, level available (where measurement was unsuccessful the number analysed is lower than the overall number analysed).
  Group 1c, 2 and 3 participants did not have a lytic bone lesion identified on novel MR scan, and were therefore not included in the analysis.
Measure: Number (95% Confidence Interval); unit: Pearson's correlation coefficient
Groups:
- Group 1a: New Myeloma: All patients with new myeloma at recruitment.
- Group 1b: Relapsed Myeloma: All patients with relapsed myeloma at recruitment.
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma
Number analyzed (Participants) | 11 | 3
Pearson's correlation coefficient
  ADC vs serum paraprotein: number analyzed (Participants) | 4 | 1
  ADC vs serum paraprotein | -0.66 [-0.99 to 0.82] | NA [NA to NA] — Only one data point, so not amenable to Pearson's correlation coefficient
  ADC vs serum paraprotein-associated immunoglobulin level: number analyzed (Participants) | 9 | 3
  ADC vs serum paraprotein-associated immunoglobulin level | -0.28 [-0.79 to 0.48] | 0.48 [NA to NA] — Only three data points, hence 95% confidence interval cannot be reliably calculated.

2. Primary Outcome: Primary Outcome 1: Quantifying Tumour Burden [Correlations With Myeloma Response Assessment and Diagnosis System (MY-RADS) Pattern of Disease]
Description: Primary Objective 1: To assess whether the novel MR protocol and exploratory bone biomarkers can improve quantification of tumour burden in patients with new or relapsed myeloma at baseline assessment, compared to paraprotein levels alone.
  Participants' baseline novel MR scan was analysed by an expert radiologist, and pattern of disease was qualitatively classified using the MY-RADS (Myeloma Response Assessment and Diagnosis System) imaging recommendations, described in Figure 2 by Messiou et. al. [1].
  This particular section analysed whether standard clinical correlate of tumour burden (serum paraprotein) differed by radiological pattern of disease (e.g., normal, focal, diffuse).
  [1] Messiou, Christina, et al. "Guidelines for acquisition, interpretation, and reporting of whole-body MRI in myeloma: myeloma response assessment and diagnosis system (MY-RADS)." Radiology 291.1 (2019): 5-13.
Time Frame: At baseline
Population: Population is all participants who had a novel MR scan at baseline with: i) available MY-RADS pattern of disease assessment; ii) available baseline serum paraprotein.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Groups:
- MY-RADS: Normal; MY-RADS: Focal; MY-RADS: Micronodular; MY-RADS: Not Determined: MY-RADS disease pattern classification, as assessed by an expert MSK Radiologist, on baseline scans
Arm/Group | MY-RADS: Normal | MY-RADS: Focal | MY-RADS: Micronodular | MY-RADS: Not Determined
Number analyzed (Participants) | 18 | 6 | 1 | 1
grams per liter (g/L) | 13.1 (9.4) | 11.7 (7.8) | 5.4 (NA) — Only one data point, hence standard deviation could not be calculated | 17.2 (NA) — Only one data point, hence standard deviation could not be calculated
Statistical Analysis 1: Comparison: MY-RADS: Normal vs MY-RADS: Focal vs MY-RADS: Micronodular; Test type: Superiority; p = 0.7343, ANOVA

3. Primary Outcome: Primary Outcome 1: Quantifying Tumour Burden (Correlations With Bone Turnover Markers)
Description: Primary Objective 1: To assess whether the novel Magnetic Resonance (MR) protocol and exploratory bone biomarkers can improve quantification of tumour burden in patients with new or relapsed myeloma at baseline assessment, compared to paraprotein levels alone.
  This section examined correlation between baseline bone biomarkers and baseline serum paraprotein in a pooled cohort of patients from Groups 1 and 2, using Spearman's Rank Correlation Coefficients.
Time Frame: At baseline
Population: Pooled cohort of patients from Groups 1 and 2 who had measured: i) available baseline serum paraprotein; ii) by baseline bone biomarkers.
Measure: Number (95% Confidence Interval); unit: Spearman's rank correlation coefficient
Groups:
- Baseline P1NP: Baseline measurements of P1NP (Procollagen type 1 N-terminal Propeptide).
- Baseline CTX-1: Baseline measurements of CTX-1 (Type I Collagen Cross-Linked C-Telopeptide).
- Baseline ALP: Baseline measurements of ALP (Alkaline Phosphatase).
- Baseline DKK1: Baseline measurements of DKK1 (Dickkopf WNT Signaling Pathway Inhibitor 1).
- Baseline Sclerostin: Baseline measurements of sclerostin.
- Baseline RANKL:OPG: Baseline measurements of the ratio between RANKL and OPG (osteoprotegerin).
Arm/Group | Baseline P1NP | Baseline CTX-1 | Baseline ALP | Baseline DKK1 | Baseline Sclerostin | Baseline RANKL:OPG
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 28 | 28
Spearman's rank correlation coefficient | 0.31 [-0.10 to 0.64] | 0.01 [-0.41 to 0.42] | -0.18 [-0.54 to 0.24] | 0.39 [0.00 to 0.68] | 0.23 [-0.17 to 0.57] | -0.02 [-0.42 to 0.38]
Statistical Analysis 1: Comparison: Baseline DKK1; Test type: Other — Correlation; p = 0.0445, Spearman's rank correlation coeffcieitn; Spearman (r) = 0.39, 95% CI 2-sided [0.00 to 0.68]

4. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss - Inter-Group Differences in Baseline Serum P1NP (Procollagen Type 1 N-terminal Propeptide)
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  This particular section analysed the inter-group difference in baseline serum P1NP (Procollagen Type 1 N-terminal Propeptide) bone turnover marker levels, in patients from Groups 1a (new myeloma), 1b (relapsed myeloma), 1c (smouldering myeloma) and 2 (MGUS).
Time Frame: At baseline
Population: All participants recruited at baseline from Groups 1 and 2 who had successful measurement of baseline serum P1NP.
Measure: Mean (Standard Deviation); unit: microgram per litre
Groups:
- Group 1a: New Myeloma: Cohort of patients recruited as new myeloma at baseline
- Group 1b: Relapsed Myeloma: Cohort of patients recruited as relapsed myeloma at baseline
- Group 1c: Smouldering Myeloma: Cohort of patients recruited as smouldering myeloma at baseline
- Group 2: MGUS: Cohort of patients recruited as MGUS at baseline
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma | Group 1c: Smouldering Myeloma | Group 2: MGUS
Number analyzed (Participants) | 14 | 11 | 15 | 13
microgram per litre | 38.6 (23.1) | 39.5 (24.0) | 39.6 (23.1) | 39.3 (23.3)
Statistical Analysis 1: Comparison: Group 1b: Relapsed Myeloma vs Group 2: MGUS; For baseline P1NP; Test type: Superiority; p = 0.0079, Kruskal-Wallis — Dunn's multiple comparisons test
Statistical Analysis 2: Comparison: Group 1a: New Myeloma vs Group 1c: Smouldering Myeloma; For baseline sclerostin; Test type: Superiority; p = 0.0482, ANOVA — Dunn's multiple comparison test

5. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss - Inter-Group Differences in Baseline Serum CTX-1 (Collagen Cross-Linked C-Telopeptide Type I)
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  This particular section analysed the inter-group difference in baseline serum CTX-1 (Collagen Cross-Linked C-Telopeptide Type I) bone turnover marker levels, in patients from Groups 1a (new myeloma), 1b (relapsed myeloma), 1c (smouldering myeloma) and 2 (MGUS).
Time Frame: At baseline
Population: All participants recruited at baseline from Groups 1 and 2 who had successful measurement of baseline serum CTX-1.
Measure: Mean (Standard Deviation); unit: microgram per litre
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma | Group 1c: Smouldering Myeloma | Group 2: MGUS
Number analyzed (Participants) | 13 | 10 | 15 | 12
microgram per litre | 0.38 (0.33) | 0.40 (0.35) | 0.39 (0.32) | 0.39 (0.32)

6. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss - Inter-Group Differences in Baseline Serum ALP (Alkaline Phosphatase)
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  This particular section analysed the inter-group difference in baseline serum ALP (Alkaline Phosphatase) bone turnover marker levels, in patients from Groups 1a (new myeloma), 1b (relapsed myeloma), 1c (smouldering myeloma) and 2 (MGUS).
Time Frame: At baseline
Population: All participants recruited at baseline from Groups 1 and 2 who had successful measurement of baseline serum ALP.
Measure: Mean (Standard Deviation); unit: international units per litre
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma | Group 1c: Smouldering Myeloma | Group 2: MGUS
Number analyzed (Participants) | 14 | 12 | 15 | 13
international units per litre | 73.8 (34.2) | 73.3 (34.9) | 72.2 (32.0) | 74.0 (33.6)

7. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss - Inter-Group Differences in Baseline Serum DKK1 (Dickkopf WNT Signaling Pathway Inhibitor 1)
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  This particular section analysed the inter-group difference in baseline serum DKK1 (Dickkopf WNT Signaling Pathway Inhibitor 1) bone turnover marker levels, in patients from Groups 1a (new myeloma), 1b (relapsed myeloma), 1c (smouldering myeloma) and 2 (MGUS).
Time Frame: At baseline
Population: All participants recruited at baseline from Groups 1 and 2 who had successful measurement of baseline serum DKK1.
Measure: Mean (Standard Deviation); unit: picogram per litre
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma | Group 1c: Smouldering Myeloma | Group 2: MGUS
Number analyzed (Participants) | 14 | 12 | 15 | 14
picogram per litre | 3963.6 (3666.8) | 4018.9 (3506.5) | 3759.2 (3175.6) | 3924.5 (3568.6)

8. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss - Inter-Group Differences in Baseline Serum Sclerostin
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  This particular section analysed the inter-group difference in baseline serum sclerostin bone turnover marker levels, in patients from Groups 1a (new myeloma), 1b (relapsed myeloma), 1c (smouldering myeloma) and 2 (MGUS).
Time Frame: At baseline
Population: All participants recruited at baseline from Groups 1 and 2 who had successful measurement of baseline serum sclerostin.
Measure: Mean (Standard Deviation); unit: picogram per litre
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma | Group 1c: Smouldering Myeloma | Group 2: MGUS
Number analyzed (Participants) | 14 | 12 | 15 | 14
picogram per litre | 168.5 (84.1) | 165.5 (85.1) | 166.9 (86.9) | 164.9 (83.6)

9. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss - Inter-Group Differences in Baseline Serum Ratio of RANKL (Receptor Activator of Nuclear Factor Kappa-Β Ligand) and OPG (Osteoprotegerin)
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  This particular section analysed the inter-group difference in baseline ratio between RANKL (Receptor Activator of Nuclear Factor Kappa-Β Ligand) and OPG (Osteoprotegerin) [calculated as RANKL (pg/L) divided by OPG (pg/L)] bone turnover marker levels, in patients from Groups 1a (new myeloma), 1b (relapsed myeloma), 1c (smouldering myeloma) and 2 (MGUS).
Time Frame: At baseline
Population: All participants recruited at baseline from Groups 1 and 2 who had successful measurement of both baseline serum RANKL and baseline serum OPG.
Measure: Mean (Standard Deviation); unit: RANKL (pg/L) to OPG (pg/L) ratio
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma | Group 1c: Smouldering Myeloma | Group 2: MGUS
Number analyzed (Participants) | 14 | 12 | 15 | 12
RANKL (pg/L) to OPG (pg/L) ratio | 0.0170 (0.0205) | 0.0176 (0.0221) | 0.0397 (0.1524) | 0.0386 (0.1494)

10. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss (Inter-Biomarker Correlations)
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  In this particular section, Spearman's rank correlation coefficient was performed to assess correlations between all pairs of bone turnover markers, measured at baseline in a pooled cohort of participants from Groups 1 and 2:
  1. P1NP (Procollagen Type 1 N-terminal Propeptide);
  2. CTX-1 (Collagen Cross-Linked C-Telopeptide Type I);
  3. ALP (Alkaline Phosphatase);
  4. DKK1 (Dickkopf WNT Signaling Pathway Inhibitor 1);
  5. Sclerostin;
  6. Ratio of RANKL (Receptor Activator of Nuclear Factor Kappa-Β Ligand) to OPG (Osteoprotegerin).
Time Frame: At baseline
Population: Pooled population of participants from Groups 1 and 2 who had bone biomarkers measured at baseline.
Measure: Number (95% Confidence Interval); unit: Spearman's rank correlation coefficient
Arm/Group | Baseline CTX-1 | Baseline ALP | Baseline DKK1 | Baseline Sclerostin | Baseline RANKL:OPG
Number analyzed (Participants) | 50 | 54 | 54 | 54 | 51
Spearman's rank correlation coefficient
  Baseline P1NP (Spearman's Rank Correlation Coefficient) | 0.70 [0.51 to 0.82] | 0.37 [0.10 to 0.58] | 0.12 [-0.16 to 0.39] | 0.22 [-0.07 to 0.47] | -0.10 [-0.37 to 0.19]
  Baseline CTX-1 (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 0 | 54 | 54 | 54 | 51
  Baseline CTX-1 (Spearman's Rank Correlation Coefficient) |  | 0.25 [-0.04 to 0.50] | 0.00 [-0.28 to 0.29] | 0.32 [0.03 to 0.55] | -0.21 [-0.47 to 0.09]
  Baseline ALP (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 0 | 0 | 54 | 54 | 51
  Baseline ALP (Spearman's Rank Correlation Coefficient) |  |  | 0.09 [-0.19 to 0.36] | -0.04 [-0.31 to 0.24] | -0.23 [-0.48 to 0.06]
  Baseline DKK1 (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 0 | 0 | 0 | 54 | 51
  Baseline DKK1 (Spearman's Rank Correlation Coefficient) |  |  |  | 0.11 [-0.16 to 0.37] | 0.13 [-0.15 to 0.39]
  Baseline Sclerostin (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 0 | 0 | 0 | 0 | 51
  Baseline Sclerostin (Spearman's Rank Correlation Coefficient) |  |  |  |  | -0.29 [-0.53 to -0.01]
  Baseline RANKL:OPG (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Primary Outcome 2: Quantifying Bone Loss [Correlations Between Bone Turnover Markers, DXA (Dual-energy X-ray Absorptiometry) and ADC (Apparent Diffusion Coefficient)]
Description: Primary Outcome 2: To assess whether the novel magnetic resonance (MR) protocol and exploratory bone turnover markers can improve quantification of bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy Of Uncertain Significance (MGUS) at baseline assessment, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone turnover markers alone.
  In this particular section, in a pooled cohort of participants from Groups 1 and 2, Spearman's rank correlation coefficients were calculated between all baseline bone turnover biomarkers and:
  1. Baseline novel MR Apparent Diffusion Coefficient (ADC) measurements;
  2. Baseline DXA (Dual-energy X-ray Absorptiometry) BMD (Bone Mineral Density) at lumbar spine (L1-4);
  2) Baseline DXA (Dual-energy X-ray Absorptiometry) BMD (Bone Mineral Density) at femoral neck.
Time Frame: At baseline
Population: Pooled population of participants from Groups 1 and 2. Where the numbers analysed are lower than the overall number of participants analysed, this reflects either failure of paired measurements for bone turnover marker and DXA and ADC, or that ADC measurements were not indicated because baseline novel MR scan did not show a lytic lesion.
Measure: Number (95% Confidence Interval); unit: Spearman's rank correlation coefficient
Arm/Group | Baseline P1NP | Baseline CTX-1 | Baseline ALP | Baseline DKK1 | Baseline Sclerostin | Baseline RANKL:OPG
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55 | 55
Spearman's rank correlation coefficient
  DXA BMD for L1-4 (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 53 | 50 | 54 | 55 | 55 | 53
  DXA BMD for L1-4 (Spearman's Rank Correlation Coefficient) | 0.02 [-0.26 to 0.29] | 0.00 [-0.29 to 0.29] | 0.16 [-0.12 to 0.41] | 0.25 [-0.03 to 0.49] | 0.54 [0.31 to 0.71] | -0.02 [-0.30 to 0.26]
  DXA BMD for Femoral Neck (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 51 | 48 | 52 | 53 | 53 | 51
  DXA BMD for Femoral Neck (Spearman's Rank Correlation Coefficient) | 0.09 [-0.20 to 0.37] | 0.14 [-0.16 to 0.41] | 0.11 [-0.17 to 0.38] | 0.19 [-0.10 to 0.44] | 0.40 [0.13 to 0.61] | 0.10 [-0.19 to 0.37]
  Novel MR ADC Measurement (Spearman's Rank Correlation Coefficient): number analyzed (Participants) | 12 | 10 | 12 | 12 | 12 | 12
  Novel MR ADC Measurement (Spearman's Rank Correlation Coefficient) | 0.09 [-0.52 to 0.64] | -0.06 [NA to NA] — Insufficient number of paired baseline CTX-1 and novel MR ADC values to enable statistical detection of Spearman's Rank correlation coefficient | -0.27 [-0.74 to 0.37] | -0.01 [-0.59 to 0.58] | -0.42 [-0.81 to 0.21] | 0.09 [-0.30 to 0.26]

12. Primary Outcome: Primary Outcome 1+2: Quantifying Tumour Burden (Total Spinal 'Hole' Volume)
Description: * This was intended as a novel end-point produced by OCMR scientists, in which high-resolution 3D imaging of the spine and pelvis are analysed for lytic lesions (holes).
  * Unfortunately, we were unable to collect data for the total spinal hole volume and total spine collapse volume at the point of novel MR scan, due to technical challenges.
Time Frame: At baseline
Population: - Unfortunately, we were unable to collect data for the total spinal hole volume and total spine collapse volume at the point of novel MR scan, due to technical challenges.
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers
Number analyzed (Participants) | 0 | 0 | 0

13. Primary Outcome: Primary Outcome 1+2: Quantifying Tumour Burden (Total Spinal 'Collapse' Volume)
Description: * This was intended as a novel end-point produced by OCMR scientists, in which high-resolution 3D imaging of the spine and pelvis are analysed for the extent of vertebral collapse.
  * Unfortunately, we were unable to collect data for the total spinal hole volume and total spine collapse volume at the point of novel magnetic resonance (MR) scan, due to technical challenges.
Time Frame: At baseline
Population: as for outcome 12
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers
Number analyzed (Participants) | 0 | 0 | 0

14. Primary Outcome: Primary Outcome 1+2: Quantifying Tumour Burden [Osteotronix Fine Structural Analysis (FSA), Trabecular Wall Thickness]
Description: * Osteotronix' fineSA® (Fine Structural Analysis, FSA) technology extracts microstructural information from Magnetic Resonance Imaging (MRI) data sets, as a correlate of trabecular wall thickness, to indicate bone remodelling. The FSA metric has been shown to correlate tightly with gold standard bone density measurements in rats [Evans et al, 2014] and human cadaveric spine specimens [Rafferty et al, 2016].
  * In this study, we had collected data during the novel MR protocol at both baseline and follow-up time points. However, we were unable to complete analysis of the FSA metrics, because of disruptions due to COVID-19, therefore the results have not been possible to report.
Time Frame: At baseline
Population: - In this study, we had collected data during the novel MR protocol at both baseline and follow-up time points. However, we were unable to complete analysis of the FSA metrics as the company we contracted to undertake this was dissolved, an alternative is not available and there is no remaining budget. Therefore the results will never be possible to report.
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Secondary Outcome 1: Detect Longitudinal Changes in Tumour Load With Therapy [MY-RADS RAC (Myeloma Response Assessment and Diagnosis System Response Assessment Classification) vs IMWG (International Myeloma Working Group) Response Group Classification]
Description: Secondary Objective 1: To assess whether the novel Magnetic Resonance (MR) protocol can improve detection of longitudinal changes in tumour burden in patients with new or relapsed myeloma during therapy, compared to the International Myeloma Working Group (IMWG) Response Group classification alone.
  This section compared two indicators of therapy response:
  1. IMWG Response Group classification [1], based on % change in serum paraprotein
  2. MY-RADS RAC (Myeloma Response Assessment and Diagnosis System Response Assessment Classification) based on expert radiologist interpretation of paired novel MR imaging, guided by Messiou et. al. criteria [2].
  Ref:
  1. https://www.myeloma.org/resource-library/international-myeloma-working-group-imwg-uniform-response-criteria-multiple
  2. Messiou, Christina, et al. "Guidelines for acquisition, interpretation, and reporting of whole-body MRI in myeloma: myeloma response assessment and diagnosis system (MY-RADS)." Radiology 291.1 (2019): 5-13.
Time Frame: Comparison between baseline and follow-up at 6 months.
Population: Participants from Group 1 who had successfully measured paired novel MR scans and serum paraproteins, between baseline and 6-month follow-up, and with a successfully graded MY-RADS RAC, and IMWG Response Group classifications.
Measure: Count of Participants; unit: Participants
Groups:
- IMWG: Relapse; IMWG: Progressive; IMWG: Stable; IMWG: Partial Response; IMWG: Very Good Partial Response; IMWG: Complete Response: IMWG classification of therapy response
Arm/Group | IMWG: Relapse | IMWG: Progressive | IMWG: Stable | IMWG: Partial Response | IMWG: Very Good Partial Response | IMWG: Complete Response
Number analyzed (Participants) | 1 | 4 | 8 | 9 | 4 | 1
Participants
  MY-RADS RAC 1: Highly likely to be responding | 0 | 0 | 0 | 2 | 3 | 0
  MY-RADS RAC 2: Likely to be responding | 0 | 1 | 0 | 4 | 0 | 0
  MY-RADS RAC 3: Stable | 1 | 3 | 8 | 3 | 1 | 1
Statistical Analysis 1: Comparison: IMWG: Relapse vs IMWG: Progressive vs IMWG: Stable vs IMWG: Partial Response vs IMWG: Very Good Partial Response vs IMWG: Complete Response; Test type: Other; p = 0.015, Fisher-Freeman-Halton exact test

16. Secondary Outcome: Secondary Outcome 1: Detect Longitudinal Changes in Tumour Load With Therapy [MY-RADS RAC (Myeloma Response Assessment and Diagnosis System Response Assessment Classification) vs % Change in ADC (Apparent Diffusion Coefficient)]
Description: Secondary Objective 1: To assess whether the novel Magnetic Resonance (MR) protocol can improve detection of longitudinal changes in tumour burden in patients with new or relapsed myeloma during therapy, compared to the International Myeloma Working Group (IMWG) Response Group classification alone.
  This section compared two indicators of therapy response:
  1. % change in Apparent Diffusion Coefficient (ADC) measurements in participants where there was a lytic bone lesion identified on both baseline and follow-up novel MR scan amenable to ADC measurement [1].
  2. MY-RADS RAC (Myeloma Response Assessment and Diagnosis System Response Assessment Classification) based on expert radiologist interpretation of paired novel MR imaging, guided by Messiou et. al. criteria [1].
  Ref:
  [1] Messiou, Christina, et al. "Guidelines for acquisition, interpretation, and reporting of whole-body MRI in myeloma: myeloma response assessment and diagnosis system (MY-RADS)." Radiology 291.1 (2019): 5-13
Time Frame: Comparison between baseline and follow-up at 6 month
Population: Participants with new or relapsed myeloma who had successfully measured paired novel MR scans at baseline and 6-month follow-up, with a successfully graded MY-RADS RAC, and a lytic bone lesion also a lytic bone lesion amenable to longitudinal calculation of % change in ADC.
Measure: Mean (Standard Deviation); unit: ADC Ratio (follow-up / baseline)
Groups:
- Group 1a: New Myeloma: Patients from Group 1a who had MY-RADS RAC score
- Group 1b: Relapsed Myeloma: Patients from Group 1b who had MY-RADS RAC score
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma
Number analyzed (Participants) | 5 | 2
ADC Ratio (follow-up / baseline)
  MY-RADS RAC 1: Highly likely to be responding: number analyzed (Participants) | 1 | 1
  MY-RADS RAC 1: Highly likely to be responding | 0.45 (NA) — 1 data point, not amenable to standard deviation calculation | 1.40 (NA) — 1 data point, not amenable to standard deviation calculation
  MY-RADS RAC 2: Likely to be responding: number analyzed (Participants) | 2 | 1
  MY-RADS RAC 2: Likely to be responding | 1.29 (0.45) | 0.57 (NA) — 1 data point, not amenable to standard deviation calculation
  MY-RADS RAC 3: Stable: number analyzed (Participants) | 2 | 0
  MY-RADS RAC 3: Stable | 1.61 (0.45) |

17. Secondary Outcome: Secondary Outcome 1: Detect Longitudinal Changes in Tumour Load With Therapy [% Change in ADC (Apparent Diffusion Coefficient) vs IMWG (International Myeloma Working Group) Response Group Classification]
Description: Secondary Objective 1: To assess whether the novel Magnetic Resonance (MR) protocol can improve detection of longitudinal changes in tumour burden in patients with new or relapsed myeloma during therapy, compared to the International Myeloma Working Group (IMWG) Response Group classification alone.
  This section compared two indicators of therapy response:
  1. IMWG Response Group classification [1], based on % change in serum paraprotein
  2. % change in Apparent Diffusion Coefficient (ADC) measurements in participants where there was a lytic bone lesion identified on both baseline and follow-up novel MR scan amenable to ADC measurement [2].
  Ref:
  1. https://www.myeloma.org/resource-library/international-myeloma-working-group-imwg-uniform-response-criteria-multiple
  2. Messiou, Christina, et al. "Guidelines for acquisition, interpretation, and reporting of whole-body MRI in myeloma: myeloma response assessment and diagnosis system (MY-RADS)." Radiology 291.1 (2019): 5-13
Time Frame: Comparison between baseline and follow-up at 6month
Population: Participants who had successfully measured paired serum paraprotein (amenable to IMWG Response Group classification) and novel MR scans (with a lytic bone lesion amenable to ADC measurement, with a successfully calculated % change in ADC) at baseline and 6-month follow-up.
Measure: Mean (Standard Deviation); unit: ADC Ratio (follow-up / baseline)
Groups:
- Group 1a: New Myeloma: Patients with new myeloma who had a lytic bone lesion amenable to longitudinal ADC measurement, and IMWG response classification.
- Group 1b: Relapsed Myeloma: Patients with relapsed myeloma who had a lytic bone lesion amenable to longitudinal ADC measurement, and IMWG response classification.
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma
Number analyzed (Participants) | 5 | 2
ADC Ratio (follow-up / baseline)
  IMWG: Progressive: number analyzed (Participants) | 1 | 0
  IMWG: Progressive | 1.6 (NA) — Single value, not amenable to calculation of standard deviation |
  IMWG: Partial Response: number analyzed (Participants) | 3 | 2
  IMWG: Partial Response | 0.90 (0.42) | 0.99 (0.59)
  IMWG: Very Good Partial Response: number analyzed (Participants) | 1 | 0
  IMWG: Very Good Partial Response | 1.9 (NA) — Single value, not amenable to calculation of standard deviation |

18. Secondary Outcome: Secondary Outcome 2: Detect Longitudinal Changes in Bone Microarchitecture With Therapy (% Change in Bone Turnover Markers)
Description: Secondary Objective 2: To assess whether the novel Magnetic Resonance (MR) protocol and exploratory bone biomarkers can improve detection of longitudinal changes in bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy of Undetermined Significance (MGUS) during therapy, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone biomarkers alone.
  This section examined whether longitudinal change in bone turnover markers differed by chemotherapy responders vs non-responders.
  * The % change in bone biomarker measurements was expressed as a ratio of follow-up / baseline of paired measurements
  * Participants were classified by International Myeloma Working Group (IMWG) Response Group classification, as responder (partial response, very good partial response or complete response) or non-responder (stable, progressive or relapse).
Time Frame: Comparison between baseline and follow-up at 6month
Population: Pooled cohort of participants from Groups 1 and 2 who had a IMWG response classification (responder vs non-responder) and paired serum bone turnover markers measured at baseline and follow-up.
Measure: Mean (Standard Deviation); unit: Ratio (follow-up divided by baseline)
Groups:
- % Change in P1NP: % Change in measurements of P1NP (Procollagen type 1 N-terminal Propeptide).
- % Change in CTX-1: % Change in measurements of CTX-1 (Type I Collagen Cross-Linked C-Telopeptide).
- % Change in ALP: % Change in measurements of ALP (Alkaline Phosphatase).
- % Change in DKK1: % Change in measurements of DKK1 (Dickkopf WNT Signaling Pathway Inhibitor 1).
- % Change in Sclerostin: % Change in measurements of sclerostin.
- % Change in RANKL:OPG: % Change in measurements of the ratio between RANKL and OPG (osteoprotegerin).
Arm/Group | % Change in P1NP | % Change in CTX-1 | % Change in ALP | % Change in DKK1 | % Change in Sclerostin | % Change in RANKL:OPG
Number analyzed (Participants) | 30 | 30 | 32 | 30 | 31 | 29
Ratio (follow-up divided by baseline)
  IMWG Responder: number analyzed (Participants) | 15 | 15 | 17 | 15 | 16 | 15
  IMWG Responder | 0.94 (0.75) | 0.89 (0.73) | 0.85 (0.22) | 0.63 (0.40) | 1.22 (0.64) | 1.09 (0.81)
  IMWG Non-Responder: number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
  IMWG Non-Responder | 0.95 (0.21) | 1.18 (0.51) | 0.98 (0.23) | 1.15 (0.59) | 1.18 (0.41) | 1.51 (1.04)
Statistical Analysis 1: Comparison: % Change in DKK1; Test type: Other; p = 0.007, Mann-Whitney test

19. Secondary Outcome: Secondary Outcome 2: Detect Longitudinal Changes in Bone Microarchitecture With Therapy (Correlations Between % Change in Bone Turnover Markers)
Description: Secondary Objective 2: To assess whether the novel Magnetic Resonance (MR) protocol and exploratory bone biomarkers can improve detection of longitudinal changes in bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy of Undetermined Significance (MGUS) during therapy, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone biomarkers alone.
  This particular section examined the correlation between longitudinal changes in bone turnover markers between one another (calculated as a ratio of follow-up measurement divided by baseline measurement). Spearman's rank correlation was performed for the longitudinal % change between different biomarkers, to assess the relationship between longitudinal changes in these measures.
Time Frame: Comparison between baseline and follow-up at 6month
Population: Pooled population of participants from Groups 1 and 2 who had paired measurements of follow-up and baseline bone turnover markers.
  For some rows, the total number of participants analysed are less than the overall number of participants analysed, due to assay failure of some bone biomarkers variably on individual samples.
Measure: Number (95% Confidence Interval); unit: Spearman's rank correlation coefficient
Arm/Group | % Change in CTX-1 | % Change in ALP | % Change in DKK1 | % Change in Sclerostin | % Change in RANKL:OPG
Number analyzed (Participants) | 40 | 43 | 44 | 43 | 49
Spearman's rank correlation coefficient
  % Change in P1NP: number analyzed (Participants) | 40 | 40 | 42 | 41 | 37
  % Change in P1NP | 0.41 [0.10 to 0.64] | 0.36 [0.05 to 0.61] | 0.12 [-0.20 to 0.41] | 0.32 [0.00 to 0.58] | 0.41 [0.09 to 0.65]
  % Change in CTX-1: number analyzed (Participants) | 0 | 40 | 40 | 39 | 35
  % Change in CTX-1 |  | 0.08 [-0.24 to 0.39] | 0.11 [-0.22 to 0.42] | 0.26 [-0.08 to 0.54] | -0.03 [-0.37 to 0.32]
  % Change in ALP: number analyzed (Participants) | 0 | 0 | 43 | 42 | 38
  % Change in ALP |  |  | 0.23 [-0.08 to 0.51] | -0.01 [-0.32 to 0.31] | -0.13 [-0.44 to 0.21]
  % Change in DKK1: number analyzed (Participants) | 0 | 0 | 0 | 43 | 39
  % Change in DKK1 |  |  |  | 0.13 [-0.18 to 0.43] | 0.14 [-0.20 to 0.44]
  % Change in Sclerostin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 39
  % Change in Sclerostin |  |  |  |  | 0.37 [0.06 to 0.62]
  % Change in RANKL:OPG: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Secondary Outcome 2: Detect Longitudinal Changes in Bone Microarchitecture With Therapy [Correlations Between % Change in Bone Turnover Markers With % Change in Bone Mineral Density (BMD) or Apparent Diffusion Coefficient (ADC)]
Description: Secondary Objective 2: To assess whether the novel Magnetic Resonance (MR) protocol and exploratory bone biomarkers can improve detection of longitudinal changes in bone loss in patients with myeloma (new, relapsed, smouldering) and Monoclonal Gammopathy of Undetermined Significance (MGUS) during therapy, compared to Dual-energy X-ray Absorptiometry (DXA) and established bone biomarkers alone.
  This section examined the correlation (using Spearman's Rank Correlation Coefficient) between longitudinal changes (expressed as a ratio of follow-up / baseline of paired measurements) in bone turnover markers and:
  1. Longitudinal changes in DXA Bone Mineral Density (BMD) at lumbar spine (L1-4) and femoral neck;
  2. Longitudinal changes in novel MR Apparent Diffusion Coefficient (ADC) measurements.
Time Frame: Comparison between baseline and follow-up at 6month
Population: Participants from Groups 1 and 2 were analysed who had a paired bone turnover marker measurements available.
  Where the number analysed for an outcome measure is lower than the overall number of participants analysed, this is due to failure of measurement of either DXA BMD or novel MR ADC, or because ADC measurement was not indicated due to lack of a lytic bone lesion identified on MR.
Measure: Number (95% Confidence Interval); unit: Spearman's rank correlation coefficient
Arm/Group | % Change in P1NP | % Change in CTX-1 | % Change in ALP | % Change in DKK1 | % Change in Sclerostin | % Change in RANKL:OPG
Number analyzed (Participants) | 41 | 40 | 42 | 43 | 42 | 38
Spearman's rank correlation coefficient
  % Change in Novel MR ADC: number analyzed (Participants) | 7 | 6 | 7 | 7 | 7 | 7
  % Change in Novel MR ADC | -0.39 [NA to NA] — Insufficient number of participants with paired ADC measurements from paired novel MR scans, to enable statistical detection of Spearman's Rank correlation coefficient | 0.31 [NA to NA] — Insufficient number of participants with paired ADC measurements from paired novel MR scans, to enable statistical detection of Spearman's Rank correlation coefficient | -0.50 [NA to NA] — Insufficient number of participants with paired ADC measurements from paired novel MR scans, to enable statistical detection of Spearman's Rank correlation coefficient | -0.32 [NA to NA] — Insufficient number of participants with paired ADC measurements from paired novel MR scans, to enable statistical detection of Spearman's Rank correlation coefficient | -0.32 [NA to NA] — Insufficient number of participants with paired ADC measurements from paired novel MR scans, to enable statistical detection of Spearman's Rank correlation coefficient | -0.14 [NA to NA] — Insufficient number of participants with paired ADC measurements from paired novel MR scans, to enable statistical detection of Spearman's Rank correlation coefficient
  % Change in DXA BMD (L1-4) | -0.12 [-0.42 to 0.21] | -0.10 [-0.41 to 0.23] | 0.02 [-0.29 to 0.33] | 0.02 [-0.29 to 0.33] | 0.24 [-0.08 to 0.51] | -0.17 [-0.48 to 0.16]
  % Change in DXA BMD (Femoral Neck): number analyzed (Participants) | 39 | 38 | 40 | 41 | 40 | 36
  % Change in DXA BMD (Femoral Neck) | -0.20 [-0.50 to 0.13] | -0.10 [-0.41 to 0.24] | -0.17 [-0.47 to 0.16] | -0.09 [-0.39 to 0.24] | 0.00 [-0.32 to 0.32] | -0.45 [-0.68 to -0.13]

21. Secondary Outcome: Secondary Objective 3: Assess Participants' Quality of Life Throughout the Study
Description: Secondary Objective 3: To assess how quality of life compares between groups and longitudinally in patients with myeloma, Monoclonal Gammopathy of Undetermined Significance (MGUS), and healthy volunteers.
  The EuroQol 5-Dimension (EQ-5D) assess the mobility, self-care, usual activities, pain/discomfort, anxiety and depression on a 5-point scale, in which a lower score represents better quality of life (1 = 'no problems', 5 = maximum problems, for each domain). The second part of the EQ-5D assess health on a scale where 100 is the best health and 0 is the worst health.
Time Frame: At baseline and six months
Population: All participants from Groups 1, 2 and 3 were invited to complete EQ5D questionnaires at baseline and 6-month follow-up visits.
  The total number of patients analysed for each EQ5D question varied slightly depending on how many responses were received from the questionnaires.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Group 1- Myeloma: Participants recruited with myeloma
- Group 2- MGUS: Participants recruited with MGUS
- Group 3- Healthy Volunteers: Participants recruited as healthy volunteers
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers
Number analyzed (Participants) | 41 | 14 | 12
Scores on a scale
  Baseline: Mobility: number analyzed (Participants) | 38 | 13 | 12
  Baseline: Mobility | 1.29 (0.46) | 1.23 (0.44) | 1.00 (0.00)
  Baseline: Self-Care: number analyzed (Participants) | 38 | 13 | 12
  Baseline: Self-Care | 1.11 (0.31) | 1.08 (0.28) | 1.00 (0.00)
  Baseline: Usual Activities: number analyzed (Participants) | 38 | 13 | 12
  Baseline: Usual Activities | 1.45 (0.65) | 1.15 (0.38) | 1.00 (0.00)
  Baseline: Pain/Discomfort: number analyzed (Participants) | 38 | 13 | 12
  Baseline: Pain/Discomfort | 1.63 (0.63) | 1.54 (0.52) | 1.08 (0.29)
  Baseline: Anxiety/Depression: number analyzed (Participants) | 38 | 13 | 12
  Baseline: Anxiety/Depression | 1.11 (0.31) | 1.08 (0.28) | 1.00 (0.00)
  Baseline: Health Score: number analyzed (Participants) | 36 | 12 | 12
  Baseline: Health Score | 72.8 (22.6) | 83.9 (7.7) | 87.9 (5.9)
  Follow-Up: Mobility: number analyzed (Participants) | 29 | 12 | 0
  Follow-Up: Mobility | 1.34 (0.48) | 1.33 (0.49) |
  Follow-Up: Self-Care: number analyzed (Participants) | 29 | 12 | 0
  Follow-Up: Self-Care | 1.07 (0.26) | 1.17 (0.39) |
  Follow-Up: Usual Activities: number analyzed (Participants) | 29 | 12 | 0
  Follow-Up: Usual Activities | 1.38 (0.49) | 1.25 (0.45) |
  Follow-Up: Pain/Discomfort: number analyzed (Participants) | 29 | 12 | 0
  Follow-Up: Pain/Discomfort | 1.59 (0.63) | 1.42 (0.51) |
  Follow-Up: Anxiety/Depression: number analyzed (Participants) | 29 | 12 | 0
  Follow-Up: Anxiety/Depression | 1.21 (0.41) | 1.08 (0.29) |
  Follow-Up: Health Score: number analyzed (Participants) | 29 | 12 | 0
  Follow-Up: Health Score | 75.1 (20.5) | 79.0 (15.6) |

22. Secondary Outcome: Secondary Outcome 4: Assess Participants' Experience of Novel Magnetic Resonance (MR) and Dual-energy X-ray Absorptiometry (DXA) Scans
Description: This questionnaire assesses the experience of the Novel Magnetic Resonance (MR) and Dual-energy X-ray Absorptiometry (DXA) scans. Answers were recorded on a 5 point Likert scale where the lower number represents a better outcome.
  Scale descriptors:
  Q1 (Overall Experience): 1 (Very comfortable)/ 2 (Comfortable)/ 3 (Neither comfortable or uncomfortable)/ 4 (Uncomfortable)/ 5 (Very uncomfortable) Q2 (Adverse Effects): 1 (YES) / 0 (NO) Q3 (Length of Time): 0 (Too short) / 1 (Just right) / 2 (Too long) Q4 (Pain/Discomfort): 1 (No Increase)/ 2 (Mild Increase)/ 3 (Moderate Increase)/ 4 (High Increase)/ 5 (Severe Increase) Q5 (Likely to Reparticipate): 0 (Extremely Unlikely) / 1 (Unlikely) / 2 (Neither Likely or Unlikely) / 3 (Likely) / 4 (Extremely Likely) Q6 (How similar to expectations): 1 (YES) / 0 (NO) Q7 (Comfort with Staff): 1 (YES) / 0 (NO)
Time Frame: At baseline and six months
Population: Baseline: all participants from Groups 1,2,3 were invited for novel MR scan, and only participants from Groups 1 and 2 were invited for DXA Follow-up: only participants from Groups 1 and 2 were invited for a novel MR scan and also a DXA.
Measure: Mean (Standard Deviation); unit: Score on a scale (see description above)
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers
Number analyzed (Participants) | 41 | 14 | 12
Score on a scale (see description above)
  Baseline novel MR scan experience: Q1 = Overall Experience: number analyzed (Participants) | 38 | 13 | 12
  Baseline novel MR scan experience: Q1 = Overall Experience | 2.10 (0.91) | 2.10 (0.93) | 2.13 (0.92)
  Baseline novel MR scan experience: Q2 = Adverse Effects: number analyzed (Participants) | 39 | 13 | 11
  Baseline novel MR scan experience: Q2 = Adverse Effects | 0.30 (0.46) | 0.31 (0.47) | 0.33 (0.47)
  Baseline novel MR scan experience: Q3 = Length of Time: number analyzed (Participants) | 37 | 12 | 10
  Baseline novel MR scan experience: Q3 = Length of Time | 1.39 (0.49) | 1.40 (0.49) | 1.40 (0.50)
  Baseline novel MR scan experience: Q4 = Pain/Discomfort: number analyzed (Participants) | 36 | 13 | 11
  Baseline novel MR scan experience: Q4 = Pain/Discomfort | 1.75 (0.86) | 1.74 (0.87) | 1.73 (0.89)
  Baseline novel MR scan experience: Q5 = How Likely to Re-participate: number analyzed (Participants) | 37 | 13 | 11
  Baseline novel MR scan experience: Q5 = How Likely to Re-participate | 3.34 (0.91) | 3.36 (0.92) | 3.34 (0.96)
  Baseline novel MR scan experience: Q6 = How Similar to Expectations: number analyzed (Participants) | 36 | 13 | 11
  Baseline novel MR scan experience: Q6 = How Similar to Expectations | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00)
  Baseline novel MR scan experience: Q7 = Comfort with Staff: number analyzed (Participants) | 37 | 13 | 11
  Baseline novel MR scan experience: Q7 = Comfort with Staff | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00)
  Follow-up novel MR scan experience: Q1 = Overall Experience: number analyzed (Participants) | 41 | 12 | 0
  Follow-up novel MR scan experience: Q1 = Overall Experience | 2.17 (1.07) | 2.20 (1.11) |
  Follow-up novel MR scan experience: Q2 = Adverse Effects: number analyzed (Participants) | 41 | 12 | 0
  Follow-up novel MR scan experience: Q2 = Adverse Effects | 0.27 (0.45) | 0.28 (0.45) |
  Follow-up novel MR scan experience: Q3 = Length of Time: number analyzed (Participants) | 41 | 9 | 0
  Follow-up novel MR scan experience: Q3 = Length of Time | 1.30 (0.46) | 1.33 (0.48) |
  Follow-up novel MR scan experience: Q4 = Pain/Discomfort: number analyzed (Participants) | 41 | 12 | 0
  Follow-up novel MR scan experience: Q4 = Pain/Discomfort | 1.44 (0.71) | 1.48 (0.82) |
  Follow-up novel MR scan experience: Q5 = How Likely to Re-participate: number analyzed (Participants) | 41 | 12 | 0
  Follow-up novel MR scan experience: Q5 = How Likely to Re-participate | 3.29 (1.05) | 3.33 (1.05) |
  Follow-up novel MR scan experience: Q6 = How Similar to Expectations: number analyzed (Participants) | 41 | 12 | 0
  Follow-up novel MR scan experience: Q6 = How Similar to Expectations | 1.00 (0.00) | 1.00 (0.00) |
  Follow-up novel MR scan experience: Q7 = Comfort with Staff: number analyzed (Participants) | 41 | 12 | 0
  Follow-up novel MR scan experience: Q7 = Comfort with Staff | 1.00 (0.00) | 0.98 (0.16) |
  Baseline DXA scan experience: Q1 = Overall Experience: number analyzed (Participants) | 40 | 13 | 0
  Baseline DXA scan experience: Q1 = Overall Experience | 1.58 (0.72) | 1.61 (0.72) |
  Baseline DXA scan experience: Q2 = Adverse Effects: number analyzed (Participants) | 40 | 13 | 0
  Baseline DXA scan experience: Q2 = Adverse Effects | 0.11 (0.32) | 0.12 (0.33) |
  Baseline DXA scan experience: Q3 = Length of Time: number analyzed (Participants) | 39 | 13 | 0
  Baseline DXA scan experience: Q3 = Length of Time | 1.00 (0.00) | 1.00 (0.00) |
  Baseline DXA scan experience: Q4 = Pain/Discomfort: number analyzed (Participants) | 40 | 12 | 0
  Baseline DXA scan experience: Q4 = Pain/Discomfort | 1.17 (0.43) | 1.16 (0.42) |
  Baseline DXA scan experience: Q5 = How Likely to Re-participate: number analyzed (Participants) | 40 | 13 | 0
  Baseline DXA scan experience: Q5 = How Likely to Re-participate | 3.51 (0.85) | 3.53 (0.83) |
  Baseline DXA scan experience: Q6 = How Similar to Expectations: number analyzed (Participants) | 38 | 13 | 0
  Baseline DXA scan experience: Q6 = How Similar to Expectations | 0.98 (0.14) | 0.98 (0.14) |
  Baseline DXA scan experience: Q7 = Comfort with Staff: number analyzed (Participants) | 39 | 13 | 0
  Baseline DXA scan experience: Q7 = Comfort with Staff | 1.00 (0.00) | 1.00 (0.00) |
  Follow-up DXA scan experience: Q1 = Overall Experience: number analyzed (Participants) | 41 | 12 | 0
  Follow-up DXA scan experience: Q1 = Overall Experience | 1.65 (0.75) | 1.71 (0.83) |
  Follow-up DXA scan experience: Q2 = Adverse Effects: number analyzed (Participants) | 41 | 12 | 0
  Follow-up DXA scan experience: Q2 = Adverse Effects | 0.09 (0.29) | 0.10 (0.30) |
  Follow-up DXA scan experience: Q3 = Length of Time: number analyzed (Participants) | 41 | 12 | 0
  Follow-up DXA scan experience: Q3 = Length of Time | 1.05 (0.21) | 1.07 (0.26) |
  Follow-up DXA scan experience: Q4 = Pain/Discomfort: number analyzed (Participants) | 41 | 12 | 0
  Follow-up DXA scan experience: Q4 = Pain/Discomfort | 1.12 (0.32) | 1.19 (0.55) |
  Follow-up DXA scan experience: Q5 = How Likely to Re-participate: number analyzed (Participants) | 41 | 12 | 0
  Follow-up DXA scan experience: Q5 = How Likely to Re-participate | 3.63 (0.85) | 3.67 (0.85) |
  Follow-up DXA scan experience: Q6 = How Similar to Expectations: number analyzed (Participants) | 41 | 12 | 0
  Follow-up DXA scan experience: Q6 = How Similar to Expectations | 1.00 (1.00) | 1.00 (0.00) |
  Follow-up DXA scan experience: Q7 = Comfort with Staff: number analyzed (Participants) | 41 | 12 | 0
  Follow-up DXA scan experience: Q7 = Comfort with Staff | 1.00 (1.00) | 0.98 (0.15) |

23. Post Hoc Outcome: Post-Hoc Analysis: Relationship Between Intercurrent Chemotherapy and Baseline Magnetic Resonance (MR) Apparent Diffusion Coefficient (ADC) Measurements
Description: We first addressed an important practical limitation of the study design. Patients with new myeloma usually commenced chemotherapy imminently after their diagnosis, typically a few months before they were able to consent for the present study. Therefore, most patients had already started chemotherapy at the point of baseline novel Magnetic Resonance (MR) scan, and had received variable durations of chemotherapy at baseline and follow-up scans. We hypothesised that this may be a potential confounding factor, as more recent chemotherapy may reduce tumour cellularity and therefore increase diffusion [and therefore Apparent Diffusion Coefficient (ADC) measurements] at lytic bone lesions.
  In this particular section, we analysed the difference between baseline ADC measurements in patients with new and relapsed myeloma, grouped by time elapsed since chemotherapy (ongoing, recent or never chemotherapy).
Time Frame: At baseline
Population: Analysis included patients from Groups 1a and 1b who had a novel MR scan at baseline, with a lytic bone lesion identified amenable to ADC measurement.
Measure: Mean (Standard Deviation); unit: s/mm^2 (ADC measurement unit)
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma
Number analyzed (Participants) | 11 | 6
s/mm^2 (ADC measurement unit)
  Baseline ADC: Ongoing Chemotherapy: number analyzed (Participants) | 9 | 3
  Baseline ADC: Ongoing Chemotherapy | 1084.5 (432.5) | 1215.3 (319.4)
  Baseline ADC: Recent (<1yr) Chemotherapy: number analyzed (Participants) | 0 | 3
  Baseline ADC: Recent (<1yr) Chemotherapy |  | 751.7 (134.8)
  Baseline ADC: Never Chemotherapy: number analyzed (Participants) | 2 | 0
  Baseline ADC: Never Chemotherapy | 547.5 (74.2) |

24. Post Hoc Outcome: Post-Hoc Analysis: Relationship Between Intercurrent Chemotherapy and Follow-Up Magnetic Resonance (MR) Apparent Diffusion Coefficient (ADC) Measurements
Description: We first addressed an important practical limitation of the study design. Patients with new myeloma usually commenced chemotherapy imminently after their diagnosis, typically a few months before they were able to consent for the present study. Therefore, most patients had already started chemotherapy at the point of baseline novel Magnetic Resonance (MR) scan, and had received variable durations of chemotherapy at baseline and follow-up scans. We hypothesised that this may be a potential confounding factor, as more recent chemotherapy may reduce tumour cellularity and therefore increase diffusion [and therefore Apparent Diffusion Coefficient (ADC) measurements] at lytic bone lesions.
  In this particular section, we analysed the difference between follow-up ADC measurements in patients with new and relapsed myeloma, grouped by time elapsed since chemotherapy (ongoing, recent or never chemotherapy).
Time Frame: At follow-up
Population: Analysis included patients from Groups 1a and 1b who had a novel MR scan at follow-up, with a lytic bone lesion identified amenable to ADC measurement.
Measure: Mean (Standard Deviation); unit: s/mm^2 (ADC measurement unit)
Arm/Group | Group 1a: New Myeloma | Group 1b: Relapsed Myeloma
Number analyzed (Participants) | 6 | 4
s/mm^2 (ADC measurement unit)
  Follow-Up ADC: Ongoing Chemotherapy: number analyzed (Participants) | 2 | 2
  Follow-Up ADC: Ongoing Chemotherapy | 1875 (205) | 1415 (968.7)
  Follow-Up ADC: Recent (<1yr) Chemotherapy: number analyzed (Participants) | 4 | 1
  Follow-Up ADC: Recent (<1yr) Chemotherapy | 1252.3 (634.7) | 900
  Follow-Up ADC: Historic Chemotherapy (>1yr): number analyzed (Participants) | 0 | 1
  Follow-Up ADC: Historic Chemotherapy (>1yr) |  | 648

ADVERSE EVENTS:
Time Frame: The intention of this study was to assess the value of disease assessment of candidate biomarkers (using DW-MRI and analysis of peripheral blood). Therefore, all-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: The intention of this study was to assess the value of disease assessment of candidate biomarkers (using DW-MRI and analysis of peripheral blood).
  Therefore, all-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Group 1- Myeloma | Group 2- MGUS | Group 3- Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
* Unable to collect data for the total spinal hole volume and total spine collapse volume at the point of novel MR scan, due to technical challenges.
* Whilst data collection is complete, there were delays in completing the analysis for Osteotronix FSA data due to disruptions with COVID-19, therefore the results have not been reported in this Study Report at time of submission. However, there is ongoing engagement with Osteotronix to complete this analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT03951220/Prot_SAP_000.pdf